CLINICAL TRIAL: NCT06519136
Title: The Effect of Reiki Therapy on Pain Severity and Quality of Life in Patients Undergoing Hemodialysis: A Follow-Up and Evaluation Study of First-Level Reiki Versus Second-Level Reiki Application
Brief Title: The Effect of Second Level Reiki on Pain Severity and Quality of Life in Patients Receiving Hemodialysis Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Sultan ÇEÇEN, Lecturer PhD, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Distance Reiki
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Hemodialysis
Keywords: Hemodialysis; Distance Reiki; Pain; Quality of life; Nursing
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The three interviewers responsible for data collection and the patients will be blinded as to which group they are in.
  According to the lists created after block randomization in the computer environment, the researcher will obtain written consent from those who agree to participate in the research. Patients in both groups will be blinded by stating that they will receive Reiki treatment remotely. In addition, until the end of the research, the group the patient is in will not be written on the data collection forms, and all three interviewers will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distance Reiki Group (Experimental): According to Usui, the second level Reiki application will be applied for 20 minutes a day between 19.00 and 21.00 in the evening for four consecutive days by the researcher who has completed his second level training, in accordance with the "Second Level Reiki Application Protocol".
  Interventions: Other: Distance Reiki
- Sham Reiki Group (Sham Comparator): It will be stated that remote energy application will be applied to the Sham Reiki group and no application will be made.
  Interventions: Other: Sham Reiki

INTERVENTIONS:
Other: Distance Reiki — According to Usui, the second level Reiki application will be applied for 20 minutes a day between 19.00 and 21.00 in the evening for four consecutive days by the researcher who has completed his second level training, in accordance with the "Second Level Reiki Application Protocol".
  Arms: Distance Reiki Group
Other: Sham Reiki — It will be stated that remote energy application will be applied to the Sham Reiki group and no application will be made.
  Arms: Sham Reiki Group

SUMMARY:
Purpose: The aim of this study is to determine the effect of 20-minute second-level Reiki application for 4 consecutive days on pain intensity and quality of life in patients receiving hemodialysis (HD) treatment and It is a comparison of the follow-up results of the first level Reiki applied within the scope of the doctoral thesis and the second level Reiki applications to be applied within the scope of this study.

Method: The study will be conducted as a pre-test-post-test, double-blind, randomized controlled trial. After obtaining Ethical Committee approval, participants in the Reiki group will receive 20-minute Reiki sessions at the second level daily from 7:00 PM to 9:00 PM for four days, while participants in the sham Reiki group will be informed that distant energy application will be performed but no actual treatment will be administered. The researcher will plan to administer second-level Reiki sessions to 8 patients daily. Throughout the study, patients in both groups will continue their routine treatments. At the beginning and three weeks after the end of the intervention, Kidney Disease Quality of Life Scale (KDQOLTM-36) scores will be collected face-to-face at HD centers, before and after the intervention Visual Analog Scale for Pain (VAS-Pain), additionally, psychodynamic responses experienced during the first and last Reiki sessions will be evaluated by three blinded assessors via telephone in both study groups.

Results: Statistical analyses of the data will be conducted using the Statistical Package for Social Sciences (Version 22.0, SPSS Inc., Chicago, IL, USA, License: Hitit University). Depending on the homogeneity of the data distribution, appropriate parametric or nonparametric tests will be performed for data evaluation.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is the chronic, progressive and irreversible loss of kidney functions associated with many causes and consists of a total of five clinical stages that require different treatment and care. The fifth of these stages is called end-stage renal disease (ESRD), and hemodialysis (HD) is offered to patients as a renal replacement treatment option unless a successful kidney transplantation occurs at this stage. Although HD treatment is a treatment option that aims to reduce mortality and morbidity rates and improve quality of life, it can also bring about different problems caused by the disease and treatment. Many physical and psychological symptoms are observed in patients receiving HD treatment, such as pain, fatigue, dyspnea, sleep problems, restless legs syndrome, itching, muscle cramps, nausea-vomiting, loss of appetite, constipation, dry skin, sexual dysfunction, anxiety, depression, and delirium. In addition, these symptoms bring about social and economic problems and negatively affect the patient's quality of life. In patients with ESRD and receiving HD treatment; The most common symptom is pain due to reasons such as accumulation of fluid and metabolic wastes, comorbid causes such as diabetes, cardiovascular and pulmonary diseases, infections, changes in the musculoskeletal system, HD procedure, carpal tunnel syndrome, and anxiety. It is known that hemodialysis patients experience moderate to severe pain, and unless the pain they experience is eliminated, the quality of life of individuals and their motivation for the continuity of treatment are negatively affected. Therefore, the importance of pain management in these patients increases considerably. The essence of effective pain management is a multidisciplinary approach and the combined use of pharmacological and non-pharmacological methods. When the studies are examined, it is seen that pharmacological and/or complementary and integrative treatment (TIT) methods are used in the management of pain in patients receiving HD treatment. In pharmacological treatment, non-opioid analgesics such as acetaminophen, topical analgesics, gabapentinoids and tricyclic antidepressants are primarily preferred. However, patients' inability to fully express their pain, their unwillingness to increase the already existing medication load, fear of addiction or side effects of the medications to be used, ethnic or cultural factors, healthcare professionals' inability to adequately evaluate pain and lack of training in pain management are among the reasons for HD patients. There are difficulties in pain management due to reasons such as the lack of a guide on pain management. For this reason, patients prefer TIT methods such as yoga, reflexology, music therapy, relaxation exercises, aromatherapy, acupressure and Reiki instead of drug treatment.

Reiki, one of the energy-based treatments that has attracted great attention from nurses among TIT methods in recent years; It provides physical, mental and emotional healing by balancing the disrupted energy flow.

While only two studies examining the effect of Reiki on pain in patients receiving HD treatment have been found in the literature, no studies investigating its effect on quality of life have been found. Reiki is a method that can be easily learned, is non-invasive, does not require special equipment, is cost-free, easy to apply, reduces the use of analgesics and has no side effects. In addition, when applied together with standard treatment, it stands out as one of the different approaches that nurses can offer to the patient in providing pain management, as it increases the quality of life by reducing the severity of pain. Based on this point, the doctoral thesis titled "The Effect of Reiki Application on Pain Intensity and Quality of Life in Patients Receiving Hemodialysis Treatment" has a mixed design; It was conducted as a pretest-posttest, double-blind, randomized controlled study and a qualitative study with individual in-depth interviews. In the study data, it was observed that first level Reiki, applied for a total of 12 sessions for 30 minutes three times a week in the first three hours of HD, reduced the severity of pain, improved mental health, and positively affected the quality of life by reducing the symptoms and problems of kidney disease. The fact that first level Reiki application takes a long time puts pressure on the practitioner, considering the other workloads of nurse practitioners, and a limited number of patients can benefit from this application.There is also a second level (distance) Reiki application in the literature that has been applied to different patient groups and examines the effect of Reiki on pain intensity. In addition, no study has been found in the literature examining the effect of second-level Reiki on pain intensity and quality of life in HD patients, nor has there been any study examining how long the effect of Reiki application lasts. Therefore, this study aims to determine the effect of 20-minute second-level Reiki application for 4 consecutive days on pain intensity and quality of life in patients receiving HD treatment and to compare the follow-up results of first-level Reiki and second-level Reiki applications.

ELIGIBILITY:
Inclusion Criteria:

* Patients who volunteered to participate in the research and received first level Reiki within the scope of the study titled "The effect of Reiki application on pain severity and quality of life in patients receiving hemodialysis treatment",
* In patients over 65 years of age, patients with a Standardized Mini Mental Test (SMMT) score of 24 points and above will be included in the sample.

Exclusion Criteria:

* Those who do not volunteer to participate in the research,
* Deceased,
* Changing the treatment center,
* Starting to receive peritoneal dialysis treatment or having renal transplantation,
* Using another complementary integrative therapy application,
* In patients over 65 years of age, patients with an SMMT value below 24 will not be included in the sample.

Ages: 28 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-12-14 (Estimated)

PRIMARY OUTCOMES:
Pain severity measurement | Day 1
  "Visual Analog Scale (VAS-Pain)" was applied to the patients in the Reiki and sham Reiki groups before and after application. In VAS-Pain, 1-3 cm is considered a "mild pain" score, 4-6 cm is considered a "moderate pain" score, and 7-10 cm is considered a "severe pain" score.
Initial quality of life measurement | Day 1
  Initial quality of life measurement, "Kidney Disease Quality of Life -KDQOLTM-36" were applied to the patients in the Reiki and sham Reiki groups. Scores in each subscale of the KDQOLTM-36 scale range from 0 to 100, with higher scores indicating better health-related quality of life.

SECONDARY OUTCOMES:
Pain severity measurement at the end of the 4th session | Day 4
  "Visual Analog Scale (VAS-Pain)" was applied to the patients in the Reiki and sham Reiki groups before and after application. In VAS-Pain, 1-3 cm is considered a "mild pain" score, 4-6 cm is considered a "moderate pain" score, and 7-10 cm is considered a "severe pain" score.
Quality of life measurement at the end of 4 week later | 4 week later
  Quality of life measurement at the end of 4 week later, "Kidney Disease Quality of Life -KDQOLTM-36" were applied to the patients in the Reiki and sham Reiki groups. Scores in each subscale of the KDQOLTM-36 scale range from 0 to 100, with higher scores indicating better health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Çeçen, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participation data will be made available for all outcome measure
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Yilmaz CK, Karakoyun A, Yurtsever S. The Effect of Distant Reiki Applied to Individuals with Extremity Amputation on Pain Level and Holistic Well-Being: A Quasi-experimental Study. Pain Manag Nurs. 2024 Apr;25(2):e87-e92. doi: 10.1016/j.pmn.2023.11.003. Epub 2023 Nov 28. PMID 38030555
- [Background] Unal N, Bektas Akpinar N, Bek D, Yurtsever S. The Effect of Reiki on Pain, Functional Status, and Holistic Well-Being in Patients With Knee Osteoarthritis: A Randomized Controlled Trial. Orthop Nurs. 2024 Mar-Apr 01;43(2):109-118. doi: 10.1097/NOR.0000000000001017. PMID 38546686
- [Derived] Cecen S, Tasci S. Impact of Reiki Levels 1 and 2 on Pain and Quality of Life Among Hemodialysis Patients: A Comparative Study. J Holist Nurs. 2025 Nov 20:8980101251393300. doi: 10.1177/08980101251393300. Online ahead of print. PMID 41264460